CLINICAL TRIAL: NCT05762679
Title: Developing Quantitative Imaging and Other Relevant Biomarkers of Myofascial Tissues for Clinical Pain Management
Brief Title: Quantifying Myofascial Dysfunction in Post-Stroke Pain
Acronym: Myofascial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); New York University (Other); George Mason University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00354876; 1R61AT012279-01 (NIH)
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Results first posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Myofascial Dysfunction
Keywords: Glycosaminoglycan; Hyaluronic acid; Post stroke shoulder pain
MeSH Terms: interventions — Diagnostic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paretic (Experimental): Subgroups:
  Low severity PSSP - defined as focal palpable nodules that may be tender on palpation with pain rating of < 5/10 when combined with the hand-behind-neck (HBN) maneuver.
  High severity PSSP - defined as focal palpable nodules that are tender on palpation, reproducing the pain, and eliciting a pain rating of >= 5/10 when combined with the hand-behind-neck (HBN) maneuver.
  Interventions: Diagnostic Test: Imaging
- Non-Paretic (Other): The non-paretic side of the same patients serves as the control.
  Interventions: Diagnostic Test: Imaging

INTERVENTIONS:
Diagnostic Test: Imaging — Phase 1 is an imaging biomarker study.

SUMMARY:
The purpose of this study is to quantify the extent of GlycosAminoGlycan/Hyaluronic Acid (GAG/HA) accumulation using T1rho (T1ρ) MRI in the paretic versus non-paretic shoulder rotator muscles, and correlate the T1ρ Magnetic Resonance Imaging (MRI) measurements with US echo texture measurements to develop a clinic-friendly tool to infer the extent of HA accumulation; and to distinguish between latent versus active Post Stroke Shoulder Pain (PSSP) using ultrasound (US) shear strain mapping of the same muscles on the paretic side compared with the non-paretic side.

DETAILED DESCRIPTION:
Shoulder pain is extremely common after stroke and occurs in 30-70% of patients. Chronic post stroke shoulder pain (PSSP) contributes to depression, interferes with motor recovery, and decreases quality of life. Although PSSP is thought to be caused by damage to the myofascial tissues around the shoulder joint, the pathophysiology of myofascial dysfunction and pain in PSSP has not been elucidated, leading to missed opportunities for early diagnosis, and variable success with pain management. The accumulation of HA in muscle and its fascia can cause myofascial dysfunction. HA is a GAG and a chief constituent of the extracellular matrix of muscle. In physiologic quantities, it functions as a lubricant and a viscoelastic shock absorber, enabling force transmission during muscle contraction and stretch. Reduced joint mobility and spasticity can result in focal accumulation and alteration of HA in muscle, leading to the development of taut bands, dysfunctional gliding of deep fascia and muscle layers, Reduced Range of Motion (ROM), and pain. Muscle HA concentrations can be imaged using T1ρ MRI, and myofascial dysfunction can be assessed using echo texture analysis and shear strain mapping on quantitative US, which may serve as useful biomarkers to elucidate the pathophysiology of myofascial dysfunction in PSSP.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Hemiparesis from Ischemic or Hemorrhagic Stroke
* 4-120 months post-stroke with Hemiparesis since the incidence and intensity of PSSP
* Show a difference of more than 10 degrees of passive ER-ROM between non-paretic and paretic shoulders with or without pain
* Able to provide informed consent and comply with testing protocols

Exclusion Criteria:

* Received treatment for spasticity with Botulinum Toxin or Intrathecal Baclofen within the past three months
* Have another neurologic condition that may affect motor response (e.g. Parkinson's disease, Amyotrophic Lateral Sclerosis (ALS), Multiple Sclerosis (MS))
* Have a contraindication to MRI (claustrophobia, magnetic pacemakers and clips)
* Have non-musculoskeletal PSSP such as only central pain or Chronic Regional Pain Syndrome (CRPS)
* Have a complicated medical condition, or significant injury to either upper limb.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Preeti Raghavan, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were enrolled at Johns Hopkins Hospital.
Pre-assignment Details: Of 46 consented participants, 42 met inclusion criteria.
Units Other Than Participants: Shoulders
Groups:
- Subjects Post-Stroke: Subjects will undergo testing on their non-paretic arm which will serve as a proxy for "healthy" control. Subjects will undergo 3 types of quantitative imaging of the pectoralis major (key internal rotator) and infraspinatus (key external rotator) muscles of both arms
Period: Overall Study
Arm/Group | Subjects Post-Stroke
Started | 42; 84 Shoulders
Paretic Low-Severity | 20; 20 Shoulders
Paretic High-Severity | 22; 22 Shoulders
Non-paretic | 42; 42 Shoulders
Completed | 40; 80 Shoulders
Not Completed | 2; 4 Shoulders
Not completed — Withdrawal by Subject | 1
Not completed — No analyzable imaging data | 1

BASELINE CHARACTERISTICS:
Population: Total of 46 participants have been consented and 42 met the eligibility criteria. out of 42 participants who finished the study, 7 lacked usable MRI or Ultrasound images and were excluded from the analysis. 35 participants have been included in the final analysis. Out of these 35, 31 have been used for MRI analysis and, 33 have been used for ultrasound analysis.
Groups:
- Paretic - Low Severity: Low severity PSSP defined as focal palpable nodules that may be tender on palpation with pain rating of < 5/10 when combined with the hand-behind-neck (HBN) maneuver.
  Imaging: Phase 1 is an imaging biomarker study.
- Paretic - High Severity: High severity PSSP is defined as focal palpable nodules that are tender on palpation, reproducing the pain, and eliciting a pain rating of >= 5/10 when combined with the hand-behind-neck (HBN) maneuver.
  Imaging: Phase 1 is an imaging biomarker study.
- Total: Total of all reporting groups
Arm/Group | Paretic - Low Severity | Paretic - High Severity | Total
Number analyzed (Participants) | 22 | 24 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.59 (12.21) | 59.67 (9.56) | 59.63 (10.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 14 | 21
  Male | 15 | 10 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 20 | 24 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 14 | 22
  White | 10 | 6 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Time since stroke [Mean (Standard Deviation); unit: Months] | 49.64 (45.55) | 36.38 (32.69) | 42.72 (39.49)

OUTCOME MEASURES:

1. Primary Outcome: T1 Rho MRI Relaxation Time of Shoulder External Rotator (Milliseconds)
Description: Comparison of T1rho (T1ρ) MRI relaxation time of infraspinatus muscles on the paretic and non-paretic sides of patients with post stroke shoulder pain.
Time Frame: Baseline
Population: MRI data were collected from 31 participants to compare paretic side with non-paretic side. Four participants were excluded based on pre-specified MRI criteria not being met. Five participants were excluded from analysis based on not meeting pre-specified criteria for pain.
Measure: Mean (Standard Deviation); unit: milliseconds
Units Other Than Participants: shoulder
Groups:
- Paretic: Shoulder/side with stiffness due to Stroke.
- Non-Paretic: Healthy side/shoulder.
Arm/Group | Paretic | Non-Paretic
Number analyzed (Participants) | 31 | 31
Number analyzed (shoulder) | 31 | 31
milliseconds | 29.09 (3.02) | 27.15 (2.20)

2. Primary Outcome: T1 Rho MRI Relaxation Time of Shoulder Internal Rotator (Milliseconds)
Description: Comparison of T1rho (T1ρ) MRI relaxation time of pectoralis major muscles on paretic and non-paretic shoulders in patients with post stroke shoulder pain.
Time Frame: Baseline
Population: MRI data was collected from 31 participants to compare paretic side with non-paretic side. Four participants were excluded based on pre-specified MRI criteria not being met. Five participants were excluded from analysis based on not meeting pre-specified criteria for pain.
Measure: Mean (Standard Deviation); unit: milliseconds
Units Other Than Participants: shoulder
Arm/Group | Paretic | Non-Paretic
Number analyzed (Participants) | 31 | 31
Number analyzed (shoulder) | 31 | 31
milliseconds | 31.83 (3.54) | 30.96 (3.60)

3. Primary Outcome: Ultrasound Shear Strain Percentage Between Paretic vs. Non-paretic Muscles
Description: Comparison of ultrasound shear strain between pectoralis major and pectoralis minor muscles on the paretic and non-paretic sides in patients with post stroke shoulder pain.
Time Frame: Baseline
Population: Ultrasound data were collected from 33 participants to compare paretic side with non-paretic side. Two were excluded from analysis based on lack of image clarity. Five participants were excluded from analysis based on not meeting pre-specified criteria for pain.
Measure: Mean (Standard Deviation); unit: Shear strain percentage
Units Other Than Participants: shoulder
Arm/Group | Paretic | Non-Paretic
Number analyzed (Participants) | 33 | 33
Number analyzed (shoulder) | 33 | 33
Shear strain percentage | 46.54 (19.81) | 35.37 (13.95)

4. Primary Outcome: Ultrasound Shear Strain Percentage Between Paretic vs. Non-paretic Side in Patients With High Severity Post Stroke Shoulder Pain
Description: Comparison of ultrasound shear strain between pectoralis major and minor muscles on the paretic side compared with the non-paretic side in patients with high severity post stroke shoulder pain
Time Frame: Baseline
Population: Ultrasound data were collected from 18/33 participants with high severity PSSP to compare paretic side with non-paretic side.
Measure: Mean (Standard Deviation); unit: Shear strain percentage
Units Other Than Participants: shoulder
Groups:
- Paretic - High Severity: Paretic side with high severity PSSP. High severity PSSP defined as focal palpable nodules that may be tender on palpation with pain rating of >/= 5/10 when combined with the hand-behind-neck (HBN) maneuver on the paretic side.
- Non-paretic - High Severity: Non-paretic side in patients with high severity PSSP on the paretic side.
Arm/Group | Paretic - High Severity | Non-paretic - High Severity
Number analyzed (Participants) | 18 | 18
Number analyzed (shoulder) | 18 | 18
Shear strain percentage | 47.46 (20.76) | 35.67 (12.86)

ADVERSE EVENTS:
Time Frame: Up to 3 weeks
Arm/Group | Subjects Post-stroke
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT05762679/Prot_SAP_000.pdf